CLINICAL TRIAL: NCT00770692
Title: A Phase III Study of SEP-190 (Eszopiclone) in Patients With Insomnia
Brief Title: A Phase III Study of Eszopiclone in Patients With Insomnia (Study SEP 190-150)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 190-150
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2012-11-22 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-10

CONDITIONS: Insomnia
Keywords: insomnia; primary insomnia; insomnia associated with psychiatric or physical disorder(s)
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone; Aging

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Eszopiclone 1 mg- Elderly (Experimental)
  Interventions: Drug: Eszopiclone 1 mg- Elderly
- Eszopiclone 2 mg- Elderly (Experimental)
  Interventions: Drug: Eszopiclone 2 mg- Elderly
- Eszopiclone 2 mg- Non-elderly (Experimental)
  Interventions: Drug: Eszopiclone 2 mg- Non-elderly
- Eszopiclone 3 mg- Non-elderly (Experimental)
  Interventions: Drug: Eszopiclone 3 mg- Non-elderly

INTERVENTIONS:
Drug: Eszopiclone 1 mg- Elderly — Elderly participants: Eszopiclone 1 mg tablet and 1 tablet of placebo 2 mg daily by mouth at bedtime for 24 weeks.
  Dose escalation occurred after 4 weeks of treatment. Participants received 1 mg tablet additionally until the end of study treatment.
  Other Names: SEP-190
  Arms: Eszopiclone 1 mg- Elderly
Drug: Eszopiclone 2 mg- Elderly — Elderly participants: Eszopiclone 2 mg tablet and 1 tablet placebo 1 mg daily by mouth at bedtime for 24 weeks.
  Dose escalation occurred after 4 weeks of treatment. Participants received 1 mg placebo tablet additionally to maintain blind until the end of study treatment.
  Other Names: SEP-190
  Arms: Eszopiclone 2 mg- Elderly
Drug: Eszopiclone 3 mg- Non-elderly — Non-elderly participants: Eszopiclone 3 mg tablet and 1 tablet of placebo 2 mg daily by mouth at bedtime for 24 weeks.
  Dose escalation occurred after 4 weeks of treatment. Participants received 1 mg placebo tablet additionally to maintain blind until the end of study treatment.
  Other Names: SEP-190
  Arms: Eszopiclone 3 mg- Non-elderly
Drug: Eszopiclone 2 mg- Non-elderly — Non-elderly participants: Eszopiclone 2 mg tablet and 1 tablet of placebo 3 mg daily by mouth at bedtime for 24 weeks.
  Dose escalation occurred after 4 weeks of treatment. Participants received 1 mg tablet additionally until the end of study treatment.
  Other Names: SEP-190
  Arms: Eszopiclone 2 mg- Non-elderly

SUMMARY:
The purpose of this study is to evaluate the long-term safety of eszopiclone (2, 3 mg) in non-elderly patients with insomnia and eszopiclone (1, 2 mg) in elderly patients with insomnia.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blinded study to evaluate the long-term safety of SEP-190 (2, 3 mg) in non-elderly patients with insomnia and SEP-190 (1, 2 mg) in elderly patients with insomnia.

ELIGIBILITY:
Inclusion criteria:

1. Participants who submit written informed consent for study entry.
2. Participants aged greater than or equal to 20 and less than 85 years of age at the time of obtaining informed consent.
3. Participants diagnosed with primary insomnia based on the Diagnostic and Statistical Manual of Mental Disorders, text revision (DSM-IV-TR) Japanese version or diagnosed with insomnia associated with psychiatric or physical disorder(s).
4. Participants with both of the following conditions which are persistent for 4 weeks or longer before the start of observation period:

   * Total sleep time is less than or equal to 390 minutes for more than or equal to 3 days a week
   * Time to fall asleep taking more than or equal to 30 minutes for more than or equal to 3 days a week
5. Participants with data at least 2 consecutive days in diary entries during observation period and confirmed to meet the following two criteria:

   * Total sleep time of less than or equal to 390 minutes for more than or equal to 3 days a week
   * Time to fall asleep taking more than or equal to 30 minutes for more than or equal to 3 days a week

Exclusion criteria:

1. Participants with a present or history of the following disease specified in

   Mini-International Neuropsychiatric Interview (M.I.N.I.) Japanese version 5.0:
   * Risk of suicide
   * (Mild) manic episode
   * Post-traumatic stress disorder (PTSD)
   * Alcohol dependence and abuse
   * Drug (non-alcohol) dependence and abuse
   * Anorexia nervosa
   * Bulimia nervosa
   * Anti-social personality disorder
2. Participants with pharmacologically induced insomnia (drug-induced insomnia).
3. Participants with comorbid primary sleep disorders (circadian rhythm disorder, restless legs movement syndrome, periodic limb movement disorder, sleep apnea syndrome, etc.) other than primary insomnia.
4. Participants with symptoms that significantly disturb sleep such as pain, fever, diarrhea, frequent micturation, and cough.
5. Participants with unstable primary disease presenting insomnia during 4 weeks before the start of observation period.
6. Participants with organic mental disorder.

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2008-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atsushi Kamijo, Study Director — New Product Development Department, Clinical Research Center
Locations (34):
- Japan (34):
  - Nagoya, Aichi-ken
  - Akita, Akita
  - Fukuoka, Fukuoka
  - Iizuka, Fukuoka
  - Kitakyushu, Fukuoka
  - Koga, Fukuoka
  - Kurume, Fukuoka
  - Maebashi, Gunma
  - Sapporo, Hokkaido
  - Itami, Hyōgo
  - Yokohama, Kanagawa
  - Yokoyama, Kanagawa
  - Kochi, Kochi
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Kashiba, Nara
  - Urazoe, Okinawa
  - Ibaraki, Osaka
  - Kishiwada, Osaka
  - Osaka, Osaka
  - Fujimi, Saitama
  - Kusatsu, Shiga
  - Arakawa-ku, Tokyo
  - Chuo-ku, Tokyo
  - Edogawa-ku, Tokyo
  - Kodaira, Tokyo
  - Koto-ku, Tokyo
  - Minato-ku, Tokyo
  - Musashino, Tokyo
  - Ōta-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Toshima-ku, Tokyo
  - Sagamihara, Yokohama

REFERENCES:
- [Derived] Uchimura N, Kamijo A, Takase T. Effects of eszopiclone on safety, subjective measures of efficacy, and quality of life in elderly and nonelderly Japanese patients with chronic insomnia, both with and without comorbid psychiatric disorders: a 24-week, randomized, double-blind study. Ann Gen Psychiatry. 2012 Jun 25;11(1):15. doi: 10.1186/1744-859X-11-15. PMID 22731653

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 181 non-elderly & 188 elderly participants were enrolled in the screening period 1 week prior to the first dose. Among these, 20 non-elderly & 24 elderly participants discontinued during the screening period. 161 non-elderly and 164 elderly participants enrolled. 1 elderly participant enrolled for treatment did not receive treatment.
Period: Overall Study
Arm/Group | Eszopiclone 1 mg- Elderly | Eszopiclone 2 mg- Elderly | Eszopiclone 2 mg- Non-elderly | Eszopiclone 3 mg- Non-elderly
Started | 81 (1 participant whose compliance was unknown, was regarded as a "treatment compliance unknown") | 83 | 84 | 77
Completed | 69 | 74 | 70 | 66
Not Completed | 12 | 9 | 14 | 11
Not completed — Withdrawal by Subject | 7 | 9 | 9 | 6
Not completed — Adverse Event | 3 | 0 | 4 | 4
Not completed — Investigator judgment | 2 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eszopiclone 1 mg- Elderly | Eszopiclone 2 mg- Elderly | Eszopiclone 2 mg- Non-elderly | Eszopiclone 3 mg- Non-elderly | Total
Number analyzed (Participants) | 80 | 83 | 84 | 77 | 324
Age Continuous [Mean (Standard Deviation); unit: years] | 70.4 (4.5) | 70.7 (4.7) | 40.1 (10.8) | 41.9 (11.5) | 55.6 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 49 | 55 | 36 | 185
  Male | 35 | 34 | 29 | 41 | 139

OUTCOME MEASURES:

1. Secondary Outcome: Mean Change From Baseline In Sleep Latency
Description: Based on subjective symptoms, the participants recorded their sleep latency (the amount of time measured in minutes it takes to fall asleep) in a sleep diary questionnaire for the week preceding the start of the study treatment (the day on which the patient was enrolled in the treatment period), as well as between the day on which the study treatment started and the Week 4 visit. For pre-treatment (screening period), the representative value was calculated from the data of the 7 days preceding enrollment in the treatment period. A median of all the data between the day of enrollment in the treatment period and the day before dose escalation judgment was presented as the data of the overall period. The change was calculated as the sleep latency of the overall period assessment - sleep latency at baseline (screening period).
Time Frame: Baseline (screening period) and 4 weeks of treatment
Population: Efficacy analysis set: all of the 161 non-elderly participants who were enrolled in the treatment period. Among the 164 elderly participants who were enrolled in the treatment period, 163 (80 in the 1 mg group and 83 in the 2 mg group) were included in the efficacy set, excluding 1 participant in the 1 mg group who had no evaluable efficacy data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Eszopiclone 1 mg- Elderly | Eszopiclone 2 mg- Elderly | Eszopiclone 2 mg- Non-elderly | Eszopiclone 3 mg- Non-elderly
Number analyzed (Participants) | 80 | 83 | 84 | 77
minutes
  Baseline | 65.5 (40.5) | 70.7 (47.1) | 71.8 (53.5) | 64.0 (42.2)
  Overall Period (Change From Baseline) | -32.1 (35.6) | -37.0 (42.7) | -36.7 (51.8) | -32.8 (35.4)

2. Primary Outcome: Incidence of Adverse Events
Description: Incidence of adverse events was defined as: (number of participants with adverse events/ number of participants analyzed in the safety analysis set)*100.
  An adverse event was defined as any unwanted or untoward disease or its symptom, sign, or abnormality in laboratory parameters in a subject who receives a study drug. An adverse event does not necessarily have a causal relationship with the study drug. The investigator or subinvestigator evaluated adverse events and recorded the results in the case report form (CRF). The investigator or subinvestigator recorded all adverse events occurring after the start of study treatment in the CRF, irrespective of the causal relationship with the study drug or the study procedures. All data collected from the follow-up was recorded in CRF.
Time Frame: Up to 25 weeks (24 weeks treatment period & 1 week follow-up)
Population: Safety analysis set: All 161 non-elderly participants who were enrolled in the treatment period were included. All 164 elderly patients who were enrolled in the treatment period were included. The participant who was excluded from the efficacy analysis set was included in the safety analysis set because the participant had evaluable safety data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Eszopiclone 1 mg- Elderly | Eszopiclone 2 mg- Elderly | Eszopiclone 2 mg- Non-elderly | Eszopiclone 3 mg- Non-elderly
Number analyzed (Participants) | 81 | 83 | 84 | 77
Percentage of Participants | 81.5 | 79.5 | 82.1 | 87.0

3. Secondary Outcome: Mean Change From Baseline in Wake Time After Sleep Onset (WASO)
Description: Based on subjective symptoms, the participants recorded their WASO defined as total awakening time from falling asleep to final awakening in a sleep diary questionnaire for the week preceding the start of the study treatment (the day on which the patient was enrolled in the treatment period), as well as between the day on which the study treatment started and the Week 4 visit. For pre-treatment (screening period), the representative value was calculated from the data of the 7 days preceding enrollment in the treatment period. A median of all the data between the day of enrollment in the treatment period and the day before dose escalation judgment was presented as the data of the overall period. The change was calculated as the WASO of the overall period assessment - WASO at baseline (screening period).
Time Frame: Baseline (screening period) and 4 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Eszopiclone 1 mg- Elderly | Eszopiclone 2 mg- Elderly | Eszopiclone 2 mg- Non-elderly | Eszopiclone 3 mg- Non-elderly
Number analyzed (Participants) | 80 | 83 | 84 | 77
minutes
  Baseline | 61.6 (52.3) | 68.8 (63.0) | 53.2 (41.8) | 42.3 (40.8)
  Overall Period (Change From Baseline) | -30.8 (39.9) | -35.1 (-25.0) | -32.4 (36.9) | -23.3 (31.1)

4. Secondary Outcome: Mean Change From Baseline in Total Sleep Time
Description: Based on subjective symptoms, the participants recorded their total sleep time defined as total sleeping time from bedtime to final awakening in a sleep diary questionnaire for the week preceding the start of the study treatment (the day on which the patient was enrolled in the treatment period), as well as between the day on which the study treatment started and the Week 4 visit. For pre-treatment (screening period), the representative value was calculated from the data of the 7 days preceding enrollment in the treatment period. A median of all the data between the day of enrollment in the treatment period and the day before dose escalation judgment was presented as the data of the overall period. The change was calculated as the total sleep time of the overall period assessment - total sleep time at baseline (screening period).
Time Frame: Baseline (screening period) and 4 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Eszopiclone 1 mg- Elderly | Eszopiclone 2 mg- Elderly | Eszopiclone 2 mg- Non-elderly | Eszopiclone 3 mg- Non-elderly
Number analyzed (Participants) | 80 | 83 | 84 | 77
minutes
  Baseline | 314.2 (73.2) | 307.9 (60.0) | 290.7 (44.0) | 308.2 (57.7)
  Overall Period (Change From Baseline) | 63.6 (64.1) | 74.2 (61.4) | 70.2 (50.2) | 61.8 (54.7)

5. Secondary Outcome: Mean Change From Baseline in Total Number of Awakenings
Description: Based on subjective symptoms, the participants recorded their number of awakenings defined as total number of spontaneous awakenings from falling asleep to final awakening in a sleep diary questionnaire for the week preceding the start of the study treatment (the day on which the patient was enrolled in the treatment period), as well as between the day on which the study treatment started and the Week 4 visit. For pre-treatment (screening period), the representative value was calculated from the data of the 7 days preceding enrollment in the treatment period. A median of all the data between the day of enrollment in the treatment period and the day before dose escalation judgment was presented as the data of the overall period. The change was calculated as the total number of awakenings of the overall period assessment - total number of awakenings at baseline (screening period).
Time Frame: Baseline (screening period) and 4 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Awakenings
Arm/Group | Eszopiclone 1 mg- Elderly | Eszopiclone 2 mg- Elderly | Eszopiclone 2 mg- Non-elderly | Eszopiclone 3 mg- Non-elderly
Number analyzed (Participants) | 80 | 83 | 84 | 77
Number of Awakenings
  Baseline | 1.8 (0.9) | 1.9 (1.0) | 1.7 (0.9) | 1.6 (1.1)
  Overall Period (Change From Baseline) | -0.5 (0.7) | -0.5 (0.8) | -0.7 (0.9) | -0.7 (0.9)

ADVERSE EVENTS:
Groups:
- Eszopiclone 2 mg Elderly: Elderly participants: Eszopiclone 2 mg tablet and 1 tablet placebo 1 mg daily by mouth at bedtime for 24 weeks.
  Dose escalation occurred after 4 weeks of treatment. Participants received 1 mg placebo tablet additionally to maintain blind until the end of study treatment.
Arm/Group | Eszopiclone 2 mg- Non-elderly | Eszopiclone 3 mg- Non-elderly | Eszopiclone 1 mg- Elderly | Eszopiclone 2 mg Elderly
Serious Adverse Events (participants affected / at risk) | 2/84 | 2/77 | 3/81 | 3/83
Other Adverse Events (participants affected / at risk) | 69/84 | 67/77 | 66/81 | 66/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eszopiclone 2 mg- Non-elderly (N=84) | Eszopiclone 3 mg- Non-elderly (N=77) | Eszopiclone 1 mg- Elderly (N=81) | Eszopiclone 2 mg Elderly (N=83)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heat illness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eszopiclone 2 mg- Non-elderly (N=84) | Eszopiclone 3 mg- Non-elderly (N=77) | Eszopiclone 1 mg- Elderly (N=81) | Eszopiclone 2 mg Elderly (N=83)
Dysgeusia (Nervous system disorders) | 36 | 44 | 15 | 23
Nasopharyngitis (Infections and infestations) | 22 | 14 | 14 | 18
Headache (Nervous system disorders) | 3 | 1 | 4 | 5
Somnolence (Nervous system disorders) | 3 | 6 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 4 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 3
Blood creatine phosphokinase increased (Investigations) | 3 | 2 | 4 | 1
Thirst (General disorders) | 2 | 2 | 3 | 0
Glucose urine present (Investigations) | 0 | 0 | 3 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 4
Pharyngitis (Infections and infestations) | 3 | 1 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 2 | 1 | 0 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 3 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Oral Discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Reflux Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Malaise (General disorders) | 0 | 2 | 2 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 2 | 1
Cystitis (Infections and infestations) | 0 | 0 | 3 | 0
Influenza (Infections and infestations) | 0 | 0 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Alanine Aminotransferase Increased (Investigations) | 2 | 1 | 0 | 0
Blood Triglycerides Increased (Investigations) | 0 | 2 | 0 | 0
Eosinophil Count Increased (Investigations) | 2 | 0 | 0 | 0
Gamma-glutamyltransferase Increased (Investigations) | 2 | 1 | 0 | 0
White Blood Cell Count Increased (Investigations) | 1 | 2 | 2 | 1
Blood Urine Present (Investigations) | 0 | 0 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Sciatica (Nervous system disorders) | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Hypertension (Vascular disorders) | 0 | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No